CLINICAL TRIAL: NCT06213051
Title: Clinical Study to Compare the Performance of Self-collected Vaginal Samples Transported Dry to Those Transported Wet for Detection of hrHPV DNA.
Brief Title: Comparison of Self-collection Using Dry Compared to Wet Swabs for HPV Detection
Acronym: HPV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Kenya Medical Research Institute (Other); Frere Hospital, East London, South Africa (Unknown); Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: WH001
Record Dates: First submitted 2023-10-04; First posted 2024-01-19 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-10

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of sexually active adult females with an abnormal cervical cancer screening result.: Multi-center, prospective, paired, comparative diagnostic accuracy study To compare the performance of self-collected vaginal samples transported dry to those transported wet for detection of hrHPV DNA.
  Interventions:
  COPAN floq swab transported wet and dry evaluated on Roche COBAS and Cepheid Xpert HPV tests
  Interventions: Device: • COPAN Self-collection FLOQSwabs® (COPAN, Italy)

INTERVENTIONS:
Device: • COPAN Self-collection FLOQSwabs® (COPAN, Italy) — COPAN swabs evaluated on Roche COBAS and Cepheid Xpert PCRs
  Other Names: COPAN Self-collection FLOQSwabs® (COPAN, Italy) with 5ml PreservCyt Solution (Hologic)

SUMMARY:
This study will compare the performance of self-collected vaginal swabs, transported without liquid media (dry swabs) and self-collected vaginal swabs, transported in liquid media (wet swabs) for detection of hrHPV DNA LBC as the reference standard.

DETAILED DESCRIPTION:
Self-collected vaginal samples for high-risk human papillomavirus (hrHPV) DNA testing are a promising alternative cervical cancer screening method for women who are reluctant to undergo healthcare provider-collection of cervical samples. Transportation of self-collected vaginal samples using swabs stored in liquid media incur additional costs and might create testing barriers for women. Dry transport of samples has the advantage of lower cost and ease of handling. Evidence on comparisons between self-collected vaginal samples using the dry swab and those transported in liquid media is limited, particularly in low- and middle-income countries (LMICs). The effect of using dry swabs on HPV-DNA detection in LMICs needs to be determined.

This study will compare the performance of self-collected vaginal swabs, transported without liquid media (dry swabs) and self-collected vaginal swabs, transported in liquid media (wet swabs) for detection of hrHPV DNA using LBC and as reference standard.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria for participants screened and enrolled consecutively as they present at the clinical study site:

* Sexually active adult females ≥30 years of age (≥25 years of age if HIV+) presenting for treatment at a facility with an abnormal cervical cancer screening result (abnormal cytology, visual inspection with acetic acid and/or colposcopy)
* Able to understand scope of study
* Able to provide written informed consent
* Willing to provide all necessary samples

Exclusion Criteria:

* Vaccinated for HPV
* Pregnancy
* Patient not willing or unable to provide the all three swab samples (self-collected dry and wet and HCW collected cervical swabs)

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult Females only
Study Population: Participants are eligible to be included in the study only if all of the inclusion criteria and none of the exclusion criteria indicated below apply.
  Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, are not permitted.
Sampling Method: Probability Sample
Enrollment: 1306 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To compare the performance of self-collected vaginal dry swabs to self-collected vaginal wet swabs for detection of hrHPV DNA using PCR on health care provider-collected cervical samples as the reference standard. | 6 Months
  Relative sensitivity and specificity, along with the percentage difference (with 95% confidence intervals), to compare self-collected vaginal dry swabs to self-collected vaginal wet swabs for detection of hrHPV DNA using PCR as the reference standard.

SECONDARY OUTCOMES:
Compare the performance of self-collected vaginal dry swabs to provider-collected cervical samples for detection of hrHPV DNA to screen for CIN2+ lesions using LBC as the reference standard. | 6 Months
  Relative sensitivity and specificity, along with the percentage difference (with 95% confidence intervals), to compare self-collected vaginal dry swabs to provider-collected cervical samples for detection of hrHPV to screen for CIN2+ lesions using LBC on health care provider-collected cervical samples as the reference standard.
Compare the performance of self-collected vaginal wet swabs to provider-collected cervical samples for detection of hrHPV DNA to screen for CIN2+ lesions using LBC as the reference standard. | 6 Months
  Relative sensitivity and specificity, along with the percentage difference (with 95% confidence intervals), to compare self-collected vaginal wet swabs to provider-collected cervical samples for detection of hrHPV to screen for CIN2+ lesions using LBC on health care provider-collected cervical samples as the reference standard.
Compare the performance of self-collected vaginal dry swabs to self-collected vaginal wet swabs for detection of hrHPV DNA to screen for CIN2+ lesions using LBC as the reference standard. | 6 Months
  Relative sensitivity and specificity, along with the percentage difference (with 95% confidence intervals), to compare self-collected dry swabs to self-collected wet swabs for detection of hrHPV to screen for CIN2+ lesions using LBC on health care provider-collected cervical samples as the reference standard.
Assess the acceptability of self-collection vs provider-collection methods for HPV testing amongst women and health care workers. | 6 Months
  Assessment of survey responses using descriptive statistics.
Assess the usability of self-collection amongst women and to assess the usability of self-collection using vaginal dry swabs compared to self-collection using vaginal wet swabs and provider collection methods for HPV testing amongst health care workers. | 6 Months
  Assessment of survey responses using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Muriuki, Study Director — Foundation for Innovative New Diagnostics (FIND)

IPD SHARING:
Plan to Share IPD: No